CLINICAL TRIAL: NCT05840055
Title: Acceptance and Commitment Therapy with Neuromyelitis Optica Spectrum Disorder Patient and Caregiver Pilot Study
Brief Title: ACT with NMOSD Patients and Caregivers Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Collaborators: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, C. Virginia O'Hayer, Clinical Professor & Director, Jefferson Center City Clinic for Behavioral Medicine, Thomas Jefferson University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: iRISID-2023-1442
Record Dates: First submitted 2023-04-11; First posted 2023-05-03 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: NMO Spectrum Disorder
MeSH Terms: conditions — Neuromyelitis Optica | interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Acceptance and Commitment Therapy (Experimental)
  Interventions: Behavioral: Acceptance and Commitment Therapy

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy — Acceptance and Commitment Therapy is one potential intervention for reducing internalizing symptoms, increasing purpose in life, and reducing avoidance-based coping among people with NMOSD and their caregiver loved ones. ACT is a "third wave" behavioral therapy which balances encouraging life changes in the service of one's values (purpose in life) with a strong acceptance component. This novel, experiential, contextual talk therapy is an empirically supported treatment for anxiety and depression, substance use, and has proven successful in managing chronic pain, somatic problems, HIV, Pancreatic Cancer and Cystic Fibrosis.

SUMMARY:
This study will examine the effectiveness of a neuromyelitis optics spectrum disorder (NMOSD) specific Acceptance and Commitment Therapy (ACT) intervention at reducing anxiety and depression in individuals with NMOSD and their caregivers/loved ones and improving overall health outcomes in individuals with NMOSD.

DETAILED DESCRIPTION:
Neuromyelitis optica spectrum disorder (NMOSD), also known as Devic disease, is an inflammatory disorder of the central nervous system. The primary symptom of NMOSD is attacks of inflammation and damage in the optic nerves and spinal cord. Such attacks may cause rapid onset of eye pain or blindness, limb weakness, numbness, or partial paralysis, shooting pain or tingling in the neck, back or abdomen, loss of bowel and bladder control, and prolonged nausea, vomiting or hiccups. These attacks may have periods of remission and relapse, with relapses most commonly occurring years to months apart. Monophasic NMO is a less common variant of NMOSD, and is characterized by a single, severe attack that may last days or weeks. When a patient is first diagnosed with NMOSD, it is unclear whether or not they will have relapses. The psychological burden of NMOSD is documented in the empirical literature, with a focus on experience of depression, pain, sexual dysfunction, sleep issues, stigma, and impact on partners.

Between 30% and 50% of individuals with NMOSD have been found to endorse clinically significant depressive symptoms on the Beck Depression Inventory. Compared with patients with Multiple Sclerosis (MS), NMOSD patients are twice as likely to receive a formal diagnosis of Recurrent Major Depressive Disorder.

Pain, bowel and bladder dysfunction, visual impairment, reduced sexual function, and inability to work, were found to most negatively impact emotional well-being and quality of life among people with NMOSD. It is estimated that chronic pain affects over 80% of NMOSD patients, including patients without recent relapse still commonly reporting moderate or severe pain. Pain severity is the strongest negative predictor of quality of life, and the most common symptom of concern voiced by patients to their physician.

Sexual dysfunction, specifically reduced libido, decreased orgasm and erectile dysfunction have been reported by 75% of males and 75% of females living with NMOSD.

Sleep disturbance is common in NMOSD, with 64% of NMOSD patients identified as poor sleepers, with correlations with anxiety, depression, pain, disability, and disease duration. Similarly, 71.4% of NMOSD patients endorsed fatigue, with correlations with sleep disturbance, depression, pain, and quality of life.

Further contributing to the psychological burden of life with NMOSD, 60% of patients reported being affected by NMOSD-related stigma. Embarrassment due to physical limitations, perceived exclusion, avoidance/ostracism, and blame for their illness were deemed the most impactful targets of stigma.

The psychological burden is also well-defined by patients with NMOSD and their loved ones in online forums, blogs, and social media. In addition to the domains cited in the literature, patients and loved ones often discuss anxiety, delayed diagnosis, physical disability and impact on relationships as hallmark characteristics of life with NMOSD. Despite the many studies suggesting that life with NMOSD is marred by many psychological stressors, including increased depression, there does not appear to be any psychosocial intervention to date to help patients and loved ones cope with this burden. Furthermore, narratives from patients across media describe profound psychological burdens that go untreated.

Given the prevalence of depression, stress, stigma, and physical impediments associated with NMOSD, it makes sense that patients and their loved ones would resort to avoidance-based coping (distraction with television, avoiding talking about illness, avoiding reminders of illness) to manage these issues. Compared with patients with multiple sclerosis, and with healthy controls, patients with NMOSD were more likely to use mental disengagement strategies, while both NMOSD and MS patients were more likely to use acceptance and behavioral disengagement strategies, compared with healthy controls. However, while avoidance-based coping may provide an effective short-term escape from the psychological burden of NMOSD, it is considered a maladaptive coping strategy in the longer term, as avoidance can be associated with medication nonadherence, missing clinic visits, failure to inform medical providers about symptoms, and can be associated with a paradoxical increase in depression and anxiety.

While the economic burden of NMOSD, including financial cost of treatments, loss of income due to disability, and associated financial pressure on caregiver/loved ones is well known, the psychological impact of NMOSD on caregivers and loved ones remains under-studied to date. Based on PHQ-9 score, 21.1% of loved ones of NMOSD patients were found to be experiencing mild, moderate, or moderately severe depressive symptoms. However, partners did not endorse clinically significant "burden", anxiety, or depression. Rather, partners endorsed pressure to take on new roles both inside and outside of the home, during NMOSD relapses, with both male and female partners identifying challenges related to gender role shift.

Partners endorsed limiting hobbies and activities to prioritize the patient's health, particularly during a relapse, along with frustration about accommodating NMOSD symptoms in public spaces, helplessness that they cannot "fix" their partner's problems, isolation due to lack of support, and anxiety about their partner's well-being and about their own health. Male partners reported "hardly expressing thoughts and feelings about NMOSD", and reported that prior to study participation, they had "never been asked how they feel about NMOSD." Lack of caregiver support and avoidance-based coping are associated with caregiver strain and burnout. Given the physical impediments associated with NMOSD, caregivers are often responsible for managing the patient's medication regimen and transporting patients to their infusion appointments. Caregiver burnout can understandably negatively impact patient treatment engagement.

Therefore, the investigators propose a caregiver-assisted, NMOSD-specific mental health intervention. Given physical limitations associated with NMOSD, and increased comfort with telehealth over the past few years, the investigators propose a telehealth-delivered intervention will be most accessible and effective. Acceptance and Commitment Therapy is one potential intervention for reducing internalizing symptoms, increasing purpose in life, and reducing avoidance-based coping among people with NMOSD and their caregiver loved ones. ACT is a "third wave" behavioral therapy which balances encouraging life changes in the service of one's values (purpose in life) with a strong acceptance component. This novel, experiential, contextual talk therapy is an empirically supported treatment for anxiety and depression, substance use, and has proven successful in managing chronic pain, somatic problems, HIV, Pancreatic Cancer and Cystic Fibrosis.

ELIGIBILITY:
Inclusion Criteria:

* Individuals ages 18 and up with a diagnosis of NMOSD and caregiver loved ones willing to participate in the intervention.
* PHQ-9 score >4, or GAD-7 score >4
* Webcam access

Exclusion Criteria:

* History of suicidal attempts or acute suicidal ideation on clinical assessment
* Presence of psychotic disorder or symptoms
* Presence of psychiatric disorders that interfere with the participation of the study, judged by the study or treating clinician. The presence of other medical conditions that interfere with participation in the study, judged by the study or treating clinician

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-11-21 (Actual)

PRIMARY OUTCOMES:
Changes in Generalized Anxiety Disorder Questionnaire (GAD7) | Baseline, 6 weeks, and three months after study completion.
  The Generalized Anxiety Disorder Questionnaire-7 is a seven item self-report questionnaire of anxiety symptom severity, with possible scores ranging from 0-21. Higher scores indicate higher anxiety symptom severity.
Changes in Patient Health Questionnaire (PHQ-9) | Baseline, 6 weeks, and three months after study completion.
  The Patient Health Questionnaire-9 is a nine item self-report questionnaire of depression symptom severity, with possible scores ranging from 0-27. Higher scores indicate higher depression symptom severity.
Changes in Beck Anxiety Inventory (BAI) | Baseline, 6 weeks, and three months after study completion.
  The Beck Anxiety Inventory (BAI) is a widely used 21-item self-report inventory used to assess anxiety levels in adults and adolescents. Scores range from 0-63, with higher scores indicating more severe anxiety.
Changes in Beck Depression Inventory (BDI-II) | Baseline, 6 weeks, and three months after study completion.
  The Beck Depression Inventory is a 21-question multiple-choice self-report inventory, one of the most widely used psychometric tests for measuring the severity of depression. Scores range from 0-63, with higher scores indicating more severe depression.

SECONDARY OUTCOMES:
Acceptance and Action Questionnaire- version 2 (AAQ-II) | Baseline, 6 weeks, and three months after study completion.
  The Acceptance and Action Questionnaire -version 2 is a seven-item measure of acceptance and committed action, ranging from 7-49. Higher scores indicate higher psychological inflexibility, experiential avoidance, and psychological distress. Lower total scores are associated with psychological flexibility.
Cognitive Fusion Questionnaire - 13 item version | Baseline, 6 weeks, and three months after study completion.
  The Cognitive Fusion Questionnaire is a 13-item measure of cognitive fusion: rigid attachment to thoughts as truth. Total scores range from 13 - 91, with higher scores indicating a higher degree of cognitive fusion.
Brief Fatigue Inventory | 3 months prior to baseline to baseline, baseline to 3 months post-treatment
  The Brief Fatigue Inventory is a 4-item measure of self-reported fatigue - Item #4 measures the extent to which fatigue has impacted each of 6 life domains. Scores range from 0-90, with higher scores indicating higher levels of fatigue and related interference.
Telephone EDSS | Baseline, 6 weeks, and three months after study completion.
  The Telephone Assessment of the Expanded Disability Status Scale is a self-administered assessment of difficulty and interference of 8 neurologic categories associated with MS and NMOSD. Scores range from 0-10, with higher scores indicating higher degree of neurological symptoms and associated interference.
Valued Living Questionnaire | Baseline, 6 weeks, and three months after study completion.
  The Valued Living Questionnaire is a 10-item measure of how important each of 10 valued domains are to the respondent, and to what extent the respondent has been living according to these values. Possible scores range from 10-100, with higher scores indicating higher consistency in living with one's values.
EHR data re. NMOSD flares, hospitalization, appointments kept/missed | 3 months prior to baseline to baseline, baseline to 3 months post-treatment
  EHR data re. presence/absence of flares, hospitalizations, clinic visits missed/kept, infusion appts missed/delayed/kept, initiation of steroid Rx, etc.

CONTACTS AND LOCATIONS:
Locations (1):
- Thomas Jefferson University Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Esiason DC, Smith PJ, Peppers CL, Wakschal E, Andrews L, Nurse CN, Kushner HM, Drescher CF, Bruschwein H, Erler W, Hattrich T, Deshpande A, Levy M, Leist T, O'Hayer CV. ACT with NMOSD: A targeted, telehealth-delivered mental health intervention for patients & caregivers. Mult Scler Relat Disord. 2025 Oct;102:106630. doi: 10.1016/j.msard.2025.106630. Epub 2025 Jul 22. PMID 40716235